CLINICAL TRIAL: NCT06421220
Title: Clinical Efficacy and Safety Evaluation of Submucosal Injection of Indocyanine Green Tracer in 3D Fluorescent Laparoscopic Lymph Node Dissection for Gastric Cancer: a Prospective, a Multicenter, Randomized, Controlled Study Clinical Trial
Brief Title: Evaluation of the Efficacy and Safety of Indocyanine Green Tracing in 3D Fluorescent Laparoscopic Lymph Node Dissection for Gastric Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Wenbin Yu, Professor， and Chief of Gastrointestinal Surgery Department, Qilu Hospital of Shandong University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202403-012-1
Record Dates: First submitted 2024-05-13; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indocyanine green tracer 3D laparoscopic gastric cancer lymph node dissection group (Experimental)
  Interventions: Procedure: Preoperative injection of indocyanine green
- Indocyanine green tracer-free 3D laparoscopic gastric cancer lymph node dissection group (No Intervention)

INTERVENTIONS:
Procedure: Preoperative injection of indocyanine green — Submucosal injection of indocyanine green into the gastric mucosa prior to surgery， indocyanine green，25mg，powder，once
  Arms: Indocyanine green tracer 3D laparoscopic gastric cancer lymph node dissection group

SUMMARY:
Purpose of the study To evaluate whether the clinical efficacy of submucosal injection of indocyanine green tracer laparoscopic gastric cancer lymph node dissection is superior to that of laparoscopic gastric cancer lymph node dissection without indocyanine green tracer in 3D fluorescence laparoscopic mode in patients with gastric adenocarcinoma (cT1-4a, N-/+, M0). To observe the role of submucosal injection of ICG for tumor localization in fluorescence 3D fluorescence laparoscopic surgery and the application of lymph node dissection in laparoscopic radical surgery for gastric cancer.

Study design. Multicenter, randomized, open, parallel-controlled, superiority design. Subgroups Group A (experimental group): indocyanine green tracer 3D laparoscopic gastric cancer lymph node dissection group Group B (control group): no indocyanine green tracer 3D laparoscopic gastric cancer lymph node dissection group.

Study population Patients who met all the inclusion criteria and did not fall into any of the exclusion criteria were eligible to enter this study.

Randomization Patients were first evaluated preoperatively to determine that they could receive laparoscopic radical gastric cancer treatment and receive endoscopic indocyanine green labeling. Once the enrolled cases were determined to meet the admission criteria after laparoscopic exploration, they could be enrolled in this study for randomization. The central dynamic, stratified zone randomization method was used in this study, and the control factors considered were age, tumor site, and preoperative stage. Given the number of seeds and the length of the zones, SAS 9.2 programming was applied to generate the treatment allocation corresponding to the running number 484, which was deposited in the data center. A person at the participating research center was responsible for sending the enrolled case information (age, tumor site, and preoperative stage) to the randomization implementation department at the data center by email, phone, or SMS, and the contact person at each respective research center confirmed that the patient met the enrollment criteria, contacted the contact person for the assigned case in this study, and determined the enrollment of the case by further analyzing the case information, and at the same time, notified the contact person at the research center where the case was located The contact person of the research center where the case is located will be notified at the same time. Competitive enrollment was used in this study.

Blinding.

DETAILED DESCRIPTION:
Case enrollment period: complete enrollment of the required cases within 2 years.

Follow-up period: The 1st case enrollment is the starting point for follow-up, and the last case enrollment to the time of return of the postoperative pathology report (usually 2 weeks postoperatively) is the endpoint of follow-up for secondary study purposes except for the 2-year recurrence type. 2 years after the last 1 case enrollment is the follow-up endpoint for the primary study purpose.

Estimated time: 2024.5-2026.4 (completion of enrollment) - 2028.4 (completion of follow-up) Standardization of Surgical Procedures. Commonly followed principles of handling in both groups Anesthesia All surgeries were performed under general anesthesia with tracheal intubation; the use of epidural-assisted anesthesia depended on the anesthesiologist and was not prescribed in this study.

Obtaining cytologic specimens for abdominal lavage After entering the abdominal cavity, firstly, the cytology specimen of abdominal lavage was retained for postoperative examination (Specific method: ascites was taken directly when ascites was found to be present. If there is no ascites, 100 ml of saline is slowly injected into the abdominal cavity, and the washings are collected and sampled in the Douglas fossa for examination.) Intraoperative exploration After obtaining cytologic specimens from abdominal lavage, the abdominal cavity is explored to check for metastases to the liver, peritoneum, mesentery, and pelvis, and invasion of the gastric plasma membrane.

Provisions for lymph node dissection Gastric cancer D2 lymph node dissection is performed according to the Japanese Guidelines for the Treatment of Gastric Cancer (5th ed.) Lymph node dissection is performed in patients in group A. After lymph node dissection, the NIR mode is used to check for the presence of missing lymph nodes, and if there are any, remedial dissection is performed.

The rules about off-site lymph node dissection: when the tumor is located in the greater curvature of the stomach, or the splenic hilar lymph nodes are enlarged on preoperative imaging, or the lymph nodes in group 10 are visualized intraoperatively, selective splenic preservation and splenic hilar lymph node dissection will be performed for the lymph nodes in group 10; group 14 lymph nodes will also be selectively disseminated when they are visualized intraoperatively; and other off-site lymph nodes will be disseminated or not by decision of the surgeon if they are visualized intraoperatively. The cleared extrastriate lymph nodes should be sent for examination and recorded separately.

Provisions for gastrectomy According to the "Japanese Guidelines for the Treatment of Gastric Cancer" (5th edition), distal or total gastrectomy should be performed as long as the oncologic principle can be guaranteed. If the operator decides to perform total laparoscopic gastrointestinal reconstruction, a sterile marker pen is required to determine the surgical incision line based on the indocyanine green range or other methods before dissecting the gastric wall, and to preserve the photographic data.

Provision for resection of the greater omentum This study protocol requires total greater omentectomy for patients with progressive gastric cancer, and the remainder is not prescribed.

Provisions for digestive tract reconstruction The way of digestive tract reconstruction shall be decided by the surgeon according to his/her own experience and intraoperative conditions, if instrumental anastomosis is used, whether to manually reinforce the anastomosis with suture shall be decided by the surgeon, and it is not stipulated in this study protocol.

Provisions for Surgery-Related Devices and Instruments Energy devices, methods of vascular ligation, GI cutting and closing, and GI reconstruction instruments are determined by the surgeon responsible for the procedure based on experience and actual needs, and are not specified in this study protocol.

Provisions for gastric tube and abdominal drainage tube Whether to keep gastric tube or abdominal drainage tube after surgery is decided by the responsible surgeon based on experience and actual needs, and is not stipulated in this study protocol.

Provisions for other surgeries performed at the same time If intraoperative findings of comorbidities of other systems/organs are detected, and the surgeon in charge of the surgery and the consulting surgeon of the relevant department jointly decide that concurrent surgery is needed to deal with them, concurrent surgery can be performed, and the sequence is decided according to the clinical routine; however, cases are excluded from the PP set according to the exclusion criteria, and the cases are excluded from the PP set.

Provisions for the treatment of excluded cases found during surgery After the patient is judged to be a cull case by the surgeon responsible for the surgery during the operation, this study protocol is suspended, and the surgeon responsible for the surgery decides the follow-up treatment by himself/herself in accordance with the clinical practice routines of the participating centers (therapeutic decision-making on whether or not to carry out the resection of the primary gastric lesion, metastasis, etc., shall be decided by the surgeon responsible for the surgery) Provisions for laparoscopic surgery Provisions for pneumoperitoneum Carbon dioxide pneumoperitoneum is used with a maintenance pressure of 12-13 mmHg, which may be appropriately lowered in advanced age.

Provisions for poking holes and auxiliary incisions The location of puncture holes and auxiliary small incisions is not regulated, and the number of puncture holes should not exceed 5. Only 1 auxiliary small incision may be made, and it must usually be less than 10 cm. when an auxiliary small incision of more than 10 cm is required, the decision must be made at the discretion of the surgeon in charge of the procedure, and the rationale must be documented in detail in the CRF.

Definition of laparoscopic access Intra-abdominal operations must be performed using laparoscopic instruments supported by a camera system. Perigastric freeing, resection of the greater omentum, resection of the omental bursa, lymph node dissection, and management of the vasculature should be accomplished laparoscopically. Gastric resection, and digestive tract reconstruction, are permitted to be accomplished in the open state using auxiliary small incisions.

Provisions for intermediate open abdomen In the event of intraoperative intra-abdominal hemorrhage, organ injury, or other serious/life-threatening complications due to surgical manipulation, which are difficult to control laparoscopically, the abdomen must be actively staged and opened. If intraoperative complications due to carbon dioxide pneumoperitoneum occur, and the anesthesiologist and the surgeon in charge of the operation discuss that it may threaten the patient's life safety, the abdomen must be actively transferred and opened. Other technical, instrumental, and other factors that lead to an intermediate open abdomen are decided by the surgeon in charge of the operation, and the reasons are recorded. The length of the incision for a mid-rotation open abdomen was not regulated in this study. The reason for the mid-excision needs to be clearly documented in the CRF.

Follow-up of rejected cases in the laparoscopic group Whether to continue the surgery under laparoscopy or to intermediate open surgery is at the discretion of the surgeon in charge of the surgery based on clinical experience.

Technical approach to indocyanine green tracing in the study group Patients enrolled in group A (study group) were injected with 1 ml of indocyanine green (indocyanine green for injection, 25 mg/strike, indocyanine green for injection diluted to 0.625 mg/ml with sterilized water for injection) into the submucosal layer of the tumor at a total of four points in the four quadrants of the tumor before the operation, and the submucosal dark-green elevation could be observed after the injection of ICG. Intraoperative visualization of the SLN tracer was performed using ICG system products. (In cT1-2 patients, if the intraoperative position is difficult to determine, preoperative marking with a harmonized titanium clip is added).

ELIGIBILITY:
Inclusion Criteria:

Age: 18-75 years old Gastric adenocarcinoma diagnosed histopathologically by endoscopic biopsy of the primary gastric lesion (pap, tub, muc, sig, por) The preoperative clinical stage was cT1-4a, N-/+, M0, according to the AJCC-8th TNM tumor stage.

Preoperative examination did not show distant metastasis, and the tumor did not directly invade the pancreas, spleen and other adjacent organs.

Preoperative ECOG physical status score 0/1 Preoperative ASA score I-III. Patient informed consent

Exclusion Criteria:

Pregnant or nursing women Serious mental illness History of upper abdominal surgery (except history of laparoscopic cholecystectomy) History of gastric surgery (including ESD/EMR for gastric cancer) Preoperative imaging suggestive of regional fusion of enlarged lymph nodes (maximum diameter ≥3cm) History of other malignant diseases within 5 years. Neoadjuvant therapy has been implemented History of unstable angina or myocardial infarction within 6 months History of cerebral infarction or cerebral hemorrhage within 6 months History of continuous systemic corticosteroid therapy within 1 month Require concomitant surgical treatment for other diseases. Gastric cancer complications (bleeding, perforation, obstruction) requiring emergency surgery.

Pulmonary function test FEV1 <50% of the expected value Diffusely invasive gastric cancer Preoperatively confirmed tumor invading the dentate line or duodenum Previous history of iodine allergy Refusal of laparoscopic surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Estimated)
Dates: Start 2024-05-20 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
2-year disease free survival rate | 12 weeks
  Observation of the rate of disease-free survival of patients two years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Wei M, Liang Y, Wang L, Li Z, Chen Y, Yan Z, Sun D, Huang Y, Zhong X, Liu P, Yu W. Clinical Application of Indocyanine Green Fluorescence Technology in Laparoscopic Radical Gastrectomy. Front Oncol. 2022 Mar 4;12:847341. doi: 10.3389/fonc.2022.847341. eCollection 2022. PMID 35311067
- [Result] Kwon IG, Son T, Kim HI, Hyung WJ. Fluorescent Lymphography-Guided Lymphadenectomy During Robotic Radical Gastrectomy for Gastric Cancer. JAMA Surg. 2019 Feb 1;154(2):150-158. doi: 10.1001/jamasurg.2018.4267. PMID 30427990
- [Result] Kim TH, Kong SH, Park JH, Son YG, Huh YJ, Suh YS, Lee HJ, Yang HK. Assessment of the Completeness of Lymph Node Dissection Using Near-infrared Imaging with Indocyanine Green in Laparoscopic Gastrectomy for Gastric Cancer. J Gastric Cancer. 2018 Jun;18(2):161-171. doi: 10.5230/jgc.2018.18.e19. Epub 2018 Jun 28. PMID 29984066
- [Result] Lan YT, Huang KH, Chen PH, Liu CA, Lo SS, Wu CW, Shyr YM, Fang WL. A pilot study of lymph node mapping with indocyanine green in robotic gastrectomy for gastric cancer. SAGE Open Med. 2017 Aug 21;5:2050312117727444. doi: 10.1177/2050312117727444. eCollection 2017. PMID 28856007
- [Result] Huh YJ, Lee HJ, Kim TH, Choi YS, Park JH, Son YG, Suh YS, Kong SH, Yang HK. Efficacy of Assessing Intraoperative Bowel Perfusion with Near-Infrared Camera in Laparoscopic Gastric Cancer Surgery. J Laparoendosc Adv Surg Tech A. 2019 Apr;29(4):476-483. doi: 10.1089/lap.2018.0263. Epub 2018 Dec 27. PMID 30589374
- [Result] Sherwinter DA, Boni L, Bouvet M, Ferri L, Hyung WJ, Ishizawa T, Kaleya RN, Kelly K, Kokudo N, Lanzarini E, Luyer MDP, Mitsumori N, Mueller C, Park DJ, Ribero D, Rosati R, Ruurda JP, Sosef M, Schneider-Koraith S, Spinoglio G, Strong V, Takahashi N, Takeuchi H, Wijnhoven BPL, Yang HK, Dip F, Lo Menzo E, White KP, Rosenthal RJ. Use of fluorescence imaging and indocyanine green for sentinel node mapping during gastric cancer surgery: Results of an intercontinental Delphi survey. Surgery. 2022 Dec;172(6S):S29-S37. doi: 10.1016/j.surg.2022.06.036. PMID 36427927
- [Result] Chen QY, Xie JW, Zhong Q, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Tu RH, Huang ZN, Lin JL, Zheng HL, Li P, Zheng CH, Huang CM. Safety and Efficacy of Indocyanine Green Tracer-Guided Lymph Node Dissection During Laparoscopic Radical Gastrectomy in Patients With Gastric Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Apr 1;155(4):300-311. doi: 10.1001/jamasurg.2019.6033. PMID 32101269